CLINICAL TRIAL: NCT02225769
Title: Electronic Algorithms Based on Host Biomarkers Point of Care Tests to Decide on Admission and Antibiotic Prescription in Tanzanian Febrile Children
Brief Title: Electronic Algorithms Based on Host Biomarkers to Manage Febrile Children
Acronym: e-POCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Valérie D'Acremont, Group leader, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IZ01Z0_146896
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute Febrile Illness
Keywords: fever; point-of-care tests; clinical algorithms; electronic support; host biomarkers
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- e-POCT (Experimental): Febrile children managed using the e-POCT tool. The e-POCT tool is an electronic algorithm that integrates key clinical elements with the results of malaria and host biomarkers point-of-care test results (including oximetry).
  Interventions: Other: Management of febrile children using e-POCT
- ALMANACH (Active Comparator): Febrile children managed using the ALMANACH algorithm. ALMANACH is an improved Integrated Management of childhood Illness (IMCI) algorithm based on mobile phones and tablets that has already been assessed for safety and efficacy.
  Interventions: Other: Management of febrile children using ALMANACH
- Routine practice (No Intervention): Febrile children managed according to routine care such as provided by routine health facility health workers.

INTERVENTIONS:
Other: Management of febrile children using e-POCT — Use of the e-POCT tool by study clinicians for the clinical management of febrile episodes. The e-POCT tool is an electronic algorithm that integrates key clinical elements with the results of malaria and host biomarkers point-of-care test results (including oximetry).
  Arms: e-POCT
Other: Management of febrile children using ALMANACH — Management of febrile children by study clinicians using ALMANACH. ALMANACH is an improved IMCI algorithm on mobile phone or tablet
  Arms: ALMANACH

SUMMARY:
Health professionals in developing countries have limited ability to identify children at risk of dying and those in need of antibiotics. The main reasons are limited clinical skills and time, unavailability of diagnostic tests (laboratory or x-ray) and non-adherence to practice guidelines. Child mortality is therefore higher than it should be. Etiological diagnostic tests (detecting microorganisms) may not always help since the distinction between infection and disease and between mild or severe disease is not straightforward. Overprescription of antibiotics is therefore widespread and leads to the development of drug resistance. To address these challenges, decision charts for the management of febrile illness will be developed and include i) few clinical parameters simple to assess, and ii) POCTs results based on specific host markers that can discriminate between mild and severe disease, pneumonia and upper respiratory tract infections, and unspecific fevers of bacterial and of viral origin. This algorithm combining clinical and bedside laboratory tests will be built on an electronic support (android tablet). The first objective of the study is to assess the safety of new electronic decision trees that integrate simple clinical assessment and POCTs results (oxygen saturation and a combination of specific biomarkers of inflammation) as a triage tool to decide on admitting febrile children; the second objective is to assess the usefulness and safety of new electronic decision trees that integrate simple clinical assessment and POCT results (a combination of specific biomarkers of inflammation) as decision-making tool to prescribe antibiotics to non-severe febrile children. The development of such a tool will decrease mortality due to delayed admission, At the same time, it will decrease irrational use of antibiotics, and hence drug pressure and emergence of drug resistance, which represents one of the most important public health threat our world is facing today. This project has the potential of huge applicability since it is specifically designed for end-users with limited medical skills and low resources, as it is the case in most areas of developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 months and <60 months of age
* Written informed consent from the child's parent or caregiver
* Axillary temperature ≥37.5°C and/or tympanic temperature ≥38.0°C
* History of fever for ≤7 days
* First consultation for the current illness
* Live in the catchment area of the health facility

Exclusion Criteria:

* Age 60 months or greater
* Age less than 2 months
* Weight less than 2.5kg
* Chief health problem is an injury, trauma or acute poisoning

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3192 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of clinical failure by day 7 compared among the 3 study arms. | 10 months
  This outcome measure is used to compare the clinical outcome of febrile children 2-59 months of age managed using e-POCT (intervention arm), ALMANACH (reference control arm) and routine practice (routine control arm).

SECONDARY OUTCOMES:
Proportions of secondary hospitalization and death by day 30 compared among the 3 study arms. | 10 months
  This outcome measure is also used to compare the clinical outcome of febrile children 2-59 months of age managed using e-POCT (intervention arm), ALMANACH (reference control arm) and routine practice (routine control arm). This type of event is however too rare to be used as primary endpoint.
Proportions of children prescribed an antibiotic and/or antimalarial treatment at day 0 and by day 7 compared among the 3 study arms. | 10 months
  This outcome is used to compare the rational use of antimicrobials in treating febrile children using e-POCT, ALMANACH and routine care.
Proportions of children with hypoxemia, stratified by diagnostic classification (e-POCT arm) | 10 months
  The aim is to measure the proportion of febrile children with hypoxemia, stratified by diagnostic classification (e-POCT arm only).
Proportion of primarily admitted children compared among the 3 study arms. | 10 months
  The objective is to compare the performance of e-POCT, ALMANACH and routine care in identifying children at risk for life-threatening infection among febrile children.

OTHER OUTCOMES:
Diagnostic performance of combinations of host biomarkers in identifying children at risk for life-threatening infections and for clinical failure among children presenting with fever (e-POCT and ALMANACH arms). | 22 months
  The objective is to explore the performance of combinations of host biomarkers in identifying children in need for antibiotic treatment, by type of infection (ALMANACH arm).

CONTACTS AND LOCATIONS:
Overall Officials: Valérie D'Acremont, MD, PhD, MiH, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Rangi tatu, Magomeni and Tandale health centers, Dar es Salaam, Dar es Salaam Region, Tanzania

REFERENCES:
- [Derived] Laubscher F, Hartley MA, Kaiser L, Cordey S. Genomic Diversity of Torque Teno Virus in Blood Samples from Febrile Paediatric Outpatients in Tanzania: A Descriptive Cohort Study. Viruses. 2022 Jul 23;14(8):1612. doi: 10.3390/v14081612. PMID 35893678
- [Derived] Cordey S, Laubscher F, Hartley MA, Junier T, Keitel K, Docquier M, Guex N, Iseli C, Vieille G, Le Mercier P, Gleizes A, Samaka J, Mlaganile T, Kagoro F, Masimba J, Said Z, Temba H, Elbanna GH, Tapparel C, Zanella MC, Xenarios I, Fellay J, D'Acremont V, Kaiser L. Blood virosphere in febrile Tanzanian children. Emerg Microbes Infect. 2021 Dec;10(1):982-993. doi: 10.1080/22221751.2021.1925161. PMID 33929935
- [Derived] Keitel K, Samaka J, Masimba J, Temba H, Said Z, Kagoro F, Mlaganile T, Sangu W, Genton B, D'Acremont V. Safety and Efficacy of C-reactive Protein-guided Antibiotic Use to Treat Acute Respiratory Infections in Tanzanian Children: A Planned Subgroup Analysis of a Randomized Controlled Noninferiority Trial Evaluating a Novel Electronic Clinical Decision Algorithm (ePOCT). Clin Infect Dis. 2019 Nov 13;69(11):1926-1934. doi: 10.1093/cid/ciz080. PMID 30715250
- [Derived] Keitel K, Kagoro F, Samaka J, Masimba J, Said Z, Temba H, Mlaganile T, Sangu W, Rambaud-Althaus C, Gervaix A, Genton B, D'Acremont V. A novel electronic algorithm using host biomarker point-of-care tests for the management of febrile illnesses in Tanzanian children (e-POCT): A randomized, controlled non-inferiority trial. PLoS Med. 2017 Oct 23;14(10):e1002411. doi: 10.1371/journal.pmed.1002411. eCollection 2017 Oct. PMID 29059253